CLINICAL TRIAL: NCT00729391
Title: Women-Focused HIV Prevention in the Western Cape
Acronym: WC-WHC
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: Medical Research Council, South Africa (Other)
Responsible Party: Principal Investigator, Wendee Wechsberg, Principal Investigator, RTI International
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01HD058320 (NIH)
Record Dates: First submitted 2008-08-05; First posted 2008-08-07 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: HIV; Substance Abuse; Violence
Keywords: HIV; Sexual Risk; Substance Abuse; Victimization; Violence; Voluntary Counseling and Testing (VCT)
MeSH Terms: conditions — Substance-Related Disorders | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Women's CoOp
  Interventions: Behavioral: Woman-Focused Intervention (Women's Health CoOp)
- 2 (Active Comparator): Nutrition (Attention-Control)
  Interventions: Behavioral: Nutrition (Attention-Control)
- 3 (Active Comparator): Voluntary Counseling and Testing
  Interventions: Behavioral: VCT Only

INTERVENTIONS:
Behavioral: Woman-Focused Intervention (Women's Health CoOp) — Participants in this group will receive VCT and participate in two group sessions of the woman-focused intervention.
  Arms: 1
Behavioral: Nutrition (Attention-Control) — Participants in this group will receive VCT and participate in two group sessions of the nutrition intervention.
  Arms: 2
Behavioral: VCT Only — Participants in this group will receive VCT only.
  Arms: 3

SUMMARY:
The purpose of this study is to test the effectiveness of a woman-focused HIV prevention intervention combined with voluntary counseling and testing (VCT), compared to VCT only, and VCT combined with an attention-control nutrition intervention.

DETAILED DESCRIPTION:
Surveillance data indicate that HIV risk and substance use is a serious problem among South African women. This study, funded by the National Institute on Child Health and Human Development (NICHD), builds on findings from a recently completed pilot study among women in less affluent townships and communities in the Western Cape (Wechsberg et al., 2008). The pilot study tested the effectiveness of an evidence-based woman-focused intervention in reducing drug use, sexual risk, and victimization by addressing the intersection of these factors among 100 poor, substance-using women of colour.

The primary aim of this study is to test the effectiveness, through a randomized controlled trial (RCT), of VCT plus a woman-focused intervention relative to VCT only to increase knowledge and skills to reduce substance abuse, sexual risk, and victimization, and to an equal-attention (nutrition) control group at 3-, 6-, 9-, and 12-month follow-ups. A secondary aim is to examine the moderating effect of victimization (i.e., sexual and physical) and the mediating effects of HIV risk knowledge, condom use skills, sexual negotiation assertiveness, and relationship power on the effectiveness of the woman-focused groups to decrease risk related to drug use, sexual risk, and sex-related-victimization relative to the rapid testing group and to the equal-attention control group.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study, participants must be: (a) female; (b) report use of at least two drugs-alcohol, marijuana, methamphetamine (tik), Mandrax (methaqualone), cocaine (crack and/or powder), heroin (Thai White), glue, MDMA (ecstasy), or LSD-at least once a week in the past 90 days; (c) be sexually active within the past 30 days with a male partner; (d) be aged 18 to 33 years; (e) live in the communities around the airport; and (f) provide verbal consent to be screened for eligibility and written consent to participate in the study.

Exclusion Criteria:

* If participants do not meet all of the inclusion criteria, they will be excluded from the study.

Ages: 18 Years to 33 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 720 (Actual)
Dates: Start 2008-09-26 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Reduction in substance abuse, sexual risk behaviors and victimization. | Baseline, 3-month, 6-month, 9-month and 12-month

SECONDARY OUTCOMES:
The moderating effect of victimization and the mediating effects of HIV risk knowledge, condom skills, sexual negotiation assertiveness, and relationship power on the effectiveness of the woman-focused groups. | 6 and 12 month

CONTACTS AND LOCATIONS:
Locations (1):
- Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Browne FA, Wechsberg WM. The intersecting risks of substance use and HIV risk among substance-using South African men and women. Curr Opin Psychiatry. 2010 May;23(3):205-9. doi: 10.1097/YCO.0b013e32833864eb. PMID 20308902
- [Background] Wechsberg WM, Browne FA, Ellerson RM, Zule WA. Adapting the evidence-based Women's CoOp intervention to prevent human immunodeficiency virus infection in North Carolina and international settings. N C Med J. 2010 Sep-Oct;71(5):477-81. No abstract available. PMID 21473554
- [Background] Jones HE, Browne FA, Myers BJ, Carney T, Ellerson RM, Kline TL, Poulton W, Zule WA, Wechsberg WM. Pregnant and nonpregnant women in cape town, South Africa: drug use, sexual behavior, and the need for comprehensive services. Int J Pediatr. 2011;2011:353410. doi: 10.1155/2011/353410. Epub 2011 Apr 6. PMID 21541067
- [Background] Zule W, Myers B, Carney T, Novak SP, McCormick K, Wechsberg WM. Alcohol and drug use outcomes among vulnerable women living with HIV: results from the Western Cape Women's Health CoOp. AIDS Care. 2014;26(12):1494-9. doi: 10.1080/09540121.2014.933769. Epub 2014 Jul 21. PMID 25040338
- [Background] Myers B, Kline TL, Doherty IA, Carney T, Wechsberg WM. Perceived need for substance use treatment among young women from disadvantaged communities in Cape Town, South Africa. BMC Psychiatry. 2014 Apr 4;14:100. doi: 10.1186/1471-244X-14-100. PMID 24708789
- [Background] Myers B, Kline TL, Browne FA, Carney T, Parry C, Johnson K, Wechsberg WM. Ethnic differences in alcohol and drug use and related sexual risks for HIV among vulnerable women in Cape Town, South Africa: implications for interventions. BMC Public Health. 2013 Feb 26;13:174. doi: 10.1186/1471-2458-13-174. PMID 23442318
- [Background] Wechsberg WM, Myers B, Kline TL, Carney T, Browne FA, Novak SP. The Relationship of Alcohol and Other Drug Use Typologies to Sex Risk Behaviors among Vulnerable Women in Cape Town, South Africa. J AIDS Clin Res. 2012 Jul 20;S1(15):015. doi: 10.4172/2155-6113.S1-015. PMID 23403403
- [Background] Reed E, Emanuel AN, Myers B, Johnson K, Wechsberg WM. The relevance of social contexts and social action in reducing substance use and victimization among women participating in an HIV prevention intervention in Cape Town, South Africa. Subst Abuse Rehabil. 2013 Jun 28;4:55-64. doi: 10.2147/SAR.S45961. eCollection 2013. PMID 24648788
- [Background] Johnson JE, Carney T, Kline T, Browne FA, Wechsberg WM. Incarceration history relative to health, substance use, and violence in a sample of vulnerable South African women: implications for health services in criminal justice settings. Subst Abuse Rehabil. 2012 Jan 28;3(Suppl 1):59-69. doi: 10.2147/SAR.S21351. eCollection 2012. PMID 24474876
- [Background] Reed E, Myers B, Novak SP, Browne FA, Wechsberg WM. Experiences of violence and association with decreased drug abstinence among women in Cape Town, South Africa. AIDS Behav. 2015 Jan;19(1):192-8. doi: 10.1007/s10461-014-0820-1. PMID 24934652
- [Result] Wechsberg WM, Jewkes R, Novak SP, Kline T, Myers B, Browne FA, Carney T, Morgan Lopez AA, Parry C. A brief intervention for drug use, sexual risk behaviours and violence prevention with vulnerable women in South Africa: a randomised trial of the Women's Health CoOp. BMJ Open. 2013 May 28;3(5):e002622. doi: 10.1136/bmjopen-2013-002622. PMID 23793683